CLINICAL TRIAL: NCT03094026
Title: Intervention Strategies to Improve Cognitive Functioning in Hematologic Cancer Survivors After Hematopoietic Cell Transplantation
Brief Title: Cognitive Training Intervention and Attitudes Towards Genetics
Acronym: cTAG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Noha Mohamed Sharafeldin, Prinicipal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: X161221006
Record Dates: First submitted 2017-03-17; First posted 2017-03-29 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Cognitive Impairment; Hematologic Neoplasms; Hematopoietic Cell Transplant
Keywords: Hematologic cancers; Hematopoietic cell transplantation; cognitive training; genetic knowledge; genetic attitude; adult cancer survivors
MeSH Terms: conditions — Cognitive Dysfunction; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The arm will begin the Lumosity program at enrollment in the study.
  Interventions: Behavioral: Lumosity
- Wait List Control (Active Comparator): The arm will begin the Lumosity program 3 months after enrollment in the study.
  Interventions: Behavioral: Lumosity (waitlist control)

INTERVENTIONS:
Behavioral: Lumosity — Computer-based online cognitive training program using the Lumosity cognitive training program.
  Arms: Intervention
Behavioral: Lumosity (waitlist control) — Computer-based online cognitive training program using the Lumosity cognitive training program. The control group will receive the intervention after a waiting period of 12 weeks.
  Arms: Wait List Control

SUMMARY:
A pilot study to evaluate feasibility of enrollment of patients in an intervention to improve neurocognitive function in hematopoietic cell transplantation (HCT) survivors using the cognitive training Lumosity program. In addition, patients' interest in receiving information regarding genetic risk of cognitive impairment post-HCT will be measured.

DETAILED DESCRIPTION:
The investigators propose using an "off-the-shelf" product - Lumosity (http://www.lumosity.com/) - an online cognitive training program, to address the cognitive impairment in outpatient HCT survivors. The program offers over 60 tasks in game-like format that cover the main cognitive domains: processing speed, working memory, and executive function. Training will involve a daily session of 5 training tasks for 12 weeks. Each time the patient is logged in for a session, a customized report will be generated by the Lumosity program to capture performance information.

Ideally, targeting the intervention and offering it specifically to those at highest risk (integrating clinical and genetic markers) would ensure efficacy. However, evidence is lacking on whether patients are receptive to communication of individual genetic information and whether provision of such results would lead to enhanced intervention response. To realize the high expectations of personalized medicine, patients' preferences and attitudes need to be thoroughly investigated especially as more information on genetic risk becomes available. The investigators will examine patients' genetic knowledge to determine whether factual knowledge of genetics is essential for understanding genetic risk and for informing treatment decision making in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 21 years old at time of allogeneic HCT performed at UAB
* Outpatient and between 3 and 6 months post HCT
* English speaking
* Possess access to an internet-connected home computer

Exclusion criteria:

* History of pre-existing neurological disorder or documented major psychiatric disorder; significant auditory, visual, or motor impairments
* Participated in neuropsychological intervention within the past 6 months
* History of color blindness

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-21 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of HCT patients completing the 2-arm wait-listed randomized trial of cognitive training intervention for a period of 3 months | 12 weeks
  Number of participants completing the 12 week intervention
Change in cognitive function between intervention and wait list control arms from baseline to 12 weeks. | Baseline to 12 weeks
  Change in cognitive function will be measured using cognitive test scores at baseline and 12 weeks

SECONDARY OUTCOMES:
16-item survey to measure genetic factual knowledge at baseline | Baseline
  Genetic factual knowledge will be measured using a 16-item survey on knowledge about genes, chromosomes, cells, and diseases and how different characteristics are inherited from parents.
Effect size of associations of key predictors with genetic factual knowledge at baseline | Baseline
  Effect size of associations of sociodemographic characteristics such as age, gender, race/ethnicity, education and income levels with genetic factual knowledge of participants will be measured.
5 Likert scale survey questionnaire to measure importance of receiving genetic risk information | baseline
  Patient ratings will be collected on a 5 Likert scale survey questionnaire to examine importance of receiving information on genetic risk of cognitive impairment post-HCT.
5 Likert scale survey questionnaire to measure impact of receiving genetic risk information on intervention uptake | baseline
  Patient ratings will be collected on a 5 Likert scale survey questionnaire to measure association of likelihood of genetic risk of cognitive impairment (low chance vs high chance) on intervention uptake.
5 Likert scale survey questionnaire to measure impact of receiving genetic risk information on intervention adherence | baseline
  Patient ratings will be collected on a 5 Likert scale survey questionnaire to measure association of likelihood of genetic risk of cognitive impairment (low chance vs high chance) on intervention adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Noha M Sharafeldin, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No